CLINICAL TRIAL: NCT04245852
Title: Does a Video-based Education Tool Related to Strengthening Result in Different Functional Outcomes Compared to Traditional Physical Therapy Education for Patients?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic disrupted subject recruitment and primary investigator no longer with our university; no additional interest in continuing the study.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Brian Thomas Baranyi, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0007
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Patients Receiving Physical Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two groups: control group or experimental group. The control group will receive standard PT care and the experimental group will receive standard physical therapy care in addition to being provided a strength education video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will receive standard physical therapy care in addition to being provided a strength education video.
  Interventions: Other: Strength education video; Other: standard PT care
- Control Group (Active Comparator): The control group will receive standard physical therapy care at the University of Illinois at Chicago Faculty Practice.
  Interventions: Other: standard PT care

INTERVENTIONS:
Other: Strength education video — The Strength education video must be watched by the patient at the University of Illinois at Chicago Faculty Practice (UICFP) prior to leaving from the 3rd physical therapy visit. The Experimental Group (EG) will watch the video in the waiting room or other quiet available rooms on the 3rd floor within the UICFP. The video will be watched from an iPad/tablet/laptop/desktop computer device as available in the clinic. The EG will also be provided a handout with a link and quick response code to the video on YouTube.com
  Arms: Experimental group
Other: standard PT care — standard PT care

SUMMARY:
• Patients receiving physical therapy (PT) at the University of Illinois at Chicago Faculty Practice (UICFP) meeting inclusion and exclusion criteria will be randomly assigned to one of two groups: control group (CG) receiving standard care and an experimental group (EG) receiving standard care in addition to being provided a strength education video (SEV). The SEV is a short video designed to provide instructions clarifying how to do strength-based exercises by monitoring a fatigue response with a set of any exercise. The EG will watch the video with headphones in the waiting room of the UICFP on an iPad. The EG will also be provided a handout with a link and QR code to the video on YouTube.com. Functional changes with PT will be tracked for both groups using a Patient Specific Functional Scale (PSFS) questionnaire at initial evaluation, follow up at session 3 or 4, and at any date of anticipated discharge. Basic demographic data (age, sex), dates of data collection, and any discharge dates will be tracked as well. If questions arise regarding the content of the SEV then the treating physical therapist will be permitted to answer and apply the content at their discretion. All therapists will have pre-approved the content of the video to ensure there are no contradictions to their usual methods of care. Data will be gathered for up to 3 months.

DETAILED DESCRIPTION:
* Human subjects for the study will be recruited and participate in the study at the University of Illinois at Chicago Faculty Practice (UICFP) located at 1640 West Roosevelt Road, 3rd floor, Chicago IL. All of the treating physical therapists with the exception of Daniel Robinson will be participating as treating physical therapists in this study and will therefore be aware of the proceedings involved. The treating physical therapists: Aaron Keil, Brian Baranyi, Justin Payette, Deborah Davey, Benjamin Land, Richelle Caya, Amanda Montbriand, Adam Wielechowski will be screening and obtaining informed consent from study participants. Additionally, Jessica Pop will be assisting in data collection and organization of data for the study.
* Patients receiving physical therapy (PT) at the UICFP will be screened for eligibility according to inclusion and exclusion criteria by treating physical therapists including obtaining consent to participate in the study at date of initial physical therapy evaluation or before the patient leaves from the second follow up visit.

  * Checking for inclusion and exclusion criteria will be referenced by the treating therapist from the "Patient Checklist Data Form" (PCDF)
  * If a patient does not meet any of the inclusion criteria or meets one of the exclusion criteria they will be excluded from the study.
  * If a patient is being added in the above manner on a date past initial evaluation the physical therapist must record previous data needed that is available from patient records (date of evaluation, Patient Specific Functional Scale (PSFS) average score). The PSFS will be provided to all possible candidates in the clinic as part of the standard intake paperwork. Therefore, the PSFS should still be available for data after obtaining consent.
  * Upon passing exclusion and inclusion criteria and obtaining informed consent, patients will be randomized into either the control or experimental group. Only after these setup steps will the PCDF be filled out and, if appropriate, provide the Strength Education Video (SEV) for viewing.

    o Once included into the study subjects will be randomly assigned to one of two groups: control group (CG) or experimental group (EG).
  * CG will receive standard PT care
  * EG will receive standard care in addition to being provided a SEV.
* The SEV must be watched by the patient at the UICFP prior to leaving from the 3rd PT visit.
* The EG will watch the video in the waiting room or other quiet available rooms on the 3rd floor within the UICFP.
* The video will be watched from an iPad/tablet/laptop/desktop computer device as available in the clinic.
* The EG will also be provided a handout with a link and QR code to the video on YouTube.com and disclaimer from the consent form.

  * Disclaimer quoted from consent form: "Please follow the link bellow to the video hosted on YouTube.com. Please be aware that by viewing the video on YouTube.com you are agreeing to YouTube and Google's terms and conditions. This will not be sharing any of your protected health information held by the University of Illinois Hospital system or the University of Illinois at Chicago. You are not obligated to click on or view this link. It is intended as a helpful tool for your benefit. Please reach out to your treating physical therapist with any questions or concerns"
  * Treating physical therapist will record the date of SEV viewing on the PCDF. - The PCDF will be used to record patient information by the treating physical therapist and have a study subject identification (ID) number added by either Daniel Robinson or Jessica Pop when performing data entry described later in protocol.
* Subject information contained in the PCDF includes:

  * Treating Physical Therapist
  * Patient Name
  * Medical Record Number
  * Age
  * Sex
  * Subject ID code
  * Which group subject is allocated to (Control or experimental)
  * Inclusion criteria checklist
  * Exclusion criteria checklist
  * Date of evaluation
  * Evaluation PSFS score
  * Date of SEV viewing (if in EG)
  * Session number of SEV viewing (if in EG)
  * Follow up PSFS score
  * Follow up session number
  * Follow up date
  * Discharge PSFS score
  * Discharge session number
  * Discharge date
  * Secondary Discharge PSFS score
  * Secondary Discharge Session number
  * Secondary Discharge date
  * Tertiary Discharge PSFS score
  * Tertiary Discharge Session number
  * Tertiary Discharge date
  * Indication if patient was discharged early from PT or had an unplanned discharge from PT.
* PCDF sheets will be kept with physical therapists when being used to gather data or in the UICFP in a locked cabinet/drawer in the folder of the specific physical therapist separate from standard treatment notes.
* Data from the PCDF will be entered without patient names into a Private Data Excel Sheet (PDES). This spreadsheet will be kept in a Box Health Data Folder (BHDF) only available to the study investigators (Daniel Robinson, Jessica Pop, and Brian Baranyi) using a secure password containing at least: one uppercase letter, one lower case letter, one number, one symbol, and at least 8 characters.

  - Functional changes with PT will be tracked for both groups using a Patient Specific Functional Scale (PSFS) questionnaire at initial evaluation, follow up at session 3 or 4 (evaluation not counting as a session), and at any date of anticipated discharge.
* The PSFS being utilized has been altered slightly from its original form for the purpose of clarifying to patients that 10 is a high functional performance skill. This is being done due to subjective reports from clinicians that patients commonly misread the questionnaire selecting 10 as a score of low function based on pain being the common question they receive. The changes made do not involve adding any new words or content changes that would be expected to alter nature of answers.

  * If questions arise regarding the content of the SEV then the treating physical therapist will be permitted to answer and apply the content at their discretion. All therapists will have pre-approved the content of the video to ensure there are no contradictions to their usual methods of care. Data will be gathered for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving physical therapy at the University of Illinois at Chicago Faculty Practice
* Strength training is a component of the intervention plan for physical therapy

  * Strength training is being defined as any exercise aimed at improving the force production, speed, and ability of a muscle group or group of muscles by using body weight, resistance bands/cords, free weights, medicine balls, weight machines or similar equipment.

Patient consents to be part of the study prior to leaving from 3rd physical therapy (PT) clinic visit (Eval +2 sessions)

* Age 18 or older
* Has been provided a PSFS on date of initial PT evaluation

Exclusion Criteria:

* Medical History of:

  * Cancer, Fibromyalgia, Polymyositis, muscular dystrophy, Lupus, Multiple Sclerosis, Parkinson's, or any other progressive/degenerative muscle/nervous system condition, Rheumatoid arthritis
* Cognitive/psychological disorder limiting ability to comprehend educational video

  * Dementia etc.
* English not preferred language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Patient Specific Functional Scale | 3 months
  The Patient Specific Functional Scale (PSFS) is a clinical outcome tool that was designed and validated for the purpose of tracking changes in function for patients with a wide variety of clinical conditions. This is measuring up to three patient identified important activities which are each scored on a 0 to 10 scale. On this scale 0 indicates "unable to perform activity" and 10 indicates "able to perform activity"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago Physical Therapy Faculty Practice, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data. Data from this study will be compiled for research purposes but not singling out any specific participant or any participant personal identifiers (i.e. name date of birth, etc).

REFERENCES:
- See also: Please see the strength education video for the experimental group — https://youtu.be/OBEauBYGRBw